CLINICAL TRIAL: NCT01258764
Title: Series of Single Patient Trials Comparing the Efficacy Between the Most Commonly Prescribed Thiazide Diuretic in the US, Hydrochlorothiazide, and Lisinopril for the Treatment of Stage 1 Hypertension.
Brief Title: Hypertensive Ambulatory Trial to Compare the Efficacy of HCTZ and Lisinopril
Acronym: 1HAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STSI 10-5486
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension, Grade 1; Hypertension Treatment; N of 1 Study Design; Hypertension
Keywords: hypertension; Blood Pressure control; hypertension treatment; antihypertensive; N of 1 study
MeSH Terms: conditions — Hypertension; Lymphoma, Follicular | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Hydrochlorothiazide; Thiazides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisinopril (Active Comparator)
  Interventions: Drug: Lisinopril
- Hydrochlorothiazide (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Lisinopril — Lisinopril 10 mg oral, once daily for four week cycle and a 2 week cycle
  Other Names: Prinivil; Zestril; ACE inhibitor
  Arms: Lisinopril
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25 mg oral, once daily for 4 week cycle and a 2 week cycle
  Other Names: Aquazide H; Carozide; Diaqua; Esidrix; Ezide; Hydro Par; HydroDIURIL; Hydrocot; Hydrokraft; Loqua; Oretic; Thiazide; HCTZ
  Arms: Hydrochlorothiazide

SUMMARY:
The purpose of this trial is to evaluate if an objective clinical decision of anti-hypertensive therapy can be made using an N-of-1 (single patient) trial design.

DETAILED DESCRIPTION:
Personalized medicine involves choosing the optimal treatment for a patient based on data gathered by the physician that is specific to that individual. The N-of-1 or single patient trial is a study design motivated by the new era of personalized medicine. The Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7) recommends a personalized medicine approach to hypertensive drug class choice based on compelling indications. However, the hypertensive decision algorithm is limited. With the advent of new technology the amount of data available to a physician has grown substantially improving the robustness of surveying a more complete picture of the patient's health care status. Medicine is quickly becoming data intensive with new technology decreasing the cost of data collection and analysis.

The typical standard care for patients with stage 1 hypertension first involves a non-pharmacological modification of lifestyle changes. Health care providers diagnose hypertension when the blood pressure is persistently elevated after three to six visits over a several month period. JNC 7 recommends thiazide-type diuretics for Stage I hypertension for most patients. In the United States, this recommendation results in most patients being given a dose of hydrochlorothiazide (HCTZ) at 12.5 to 25 mg per day. A patient would then return for follow-up and would be prescribed a few month supply of an antihypertensive medication (e.g. HCTZ or lisinopril). The choice of treatment by the physician is based on JNC 7 guidelines, patient's risk factors, and a provider's experience.

The objective of this trial will be to evaluate if an objective clinical decision of anti-hypertensive therapy can be made using an N-of-1 (single patient) trial design. In this study we propose to do a series of N-of-1 trials in patients with stage 1 hypertension who will be randomized to alternating courses of HCTZ and lisinopril.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Grade 1 Hypertension
* Treatment naïve
* GFR > 60 within previous 3 months
* Urinary microalbumin level normal during previous 3 months

Exclusion Criteria:

* Pregnancy (Fetal morbidity and mortality may occur with the use of ACE inhibitors.)
* Uncontrolled Hyperthyroidism
* Sleep Apnea
* Primary Aldosteronism
* Renovascular Disease
* Cushing's Syndrome or steroid therapy
* No evidence of end organ damage
* EKG with evidence of LVH within previous 3 months
* Collagen Vascular Disease
* Current Smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure control defined as 24-hour ambulatory systolic and diastolic pressure average below 135/85 mmHg. | After 14 week study period with assessment of patient specific data

SECONDARY OUTCOMES:
Blood Pressure (BP) load, treatment of non-dippers, side effects, and compliance. | After 14 week study period with assessment of patient specific data
  BP load is defined as the percentage of ambulatory systolic and diastolic pressure exceeding 140 mmHg and 90 mmHg during the daytime and 120 mmHg and 80 mmHg during sleep. Systolic BP load averages 9-25% depending on age. While diastolic BP load averages 3-4%. Failure of BP to fall by at least 10 percent during sleep will define a non-dipper. Extreme dipping will be defined by a nocturnal BP decline of greater than 20 percent with a large morning increase in BP.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Patay, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Clinic, La Jolla, California, United States

REFERENCES:
- See also: Related Info — http://www.Scripps.org